CLINICAL TRIAL: NCT06805955
Title: The Effect of Hand Rehabilitation Robot on Functionality and Activities of Daily Living in Acute Stroke Rehabilitation
Brief Title: Effect of Hand Rehabilitation Robot on Acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.302-620
Record Dates: First submitted 2025-01-28; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Rehabilitation
Keywords: stroke; motor function; fine motor skills; hand robot
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurodevelopmental Group (Active Comparator): A total of 30 participants meeting inclusion criteria were divided into two groups: the Neurodevelopmental Treatment (NDT) Group (n=15) and the Hand Robot Group (n=15). Both groups completed 24 sessions over 8 weeks (3 days/week, 60 minutes/session). The NDT Group received neurodevelopmental treatment, while the Hand Robot Group received 35 minutes of NDT plus 25 minutes of hand robot-assisted therapy.The NDT program included exercises to reduce muscle tone, improve hand function, and enhance fine motor skills and daily living activities. Specific tasks involved finger and wrist movements, elbow and shoulder mobilizations, PNF exercises, and functional activities like door handle turning and zipper-pulling. Exercises were adapted to patient ability with 10 repetitions per task.Both groups received 15 minutes of electrical stimulation targeting deltoid, biceps, or forearm flexors after each session to enhance muscle strength.
  Interventions: Other: NDT
- Hand Robot Group (Experimental): In this group, participants received 25 minutes of therapy using the hand robot following neurodevelopmental treatment sessions. After the hand robot therapy, participants performed exercises designed to enhance fine motor skills. The fine motor activities included:
  Picking up buttons from one container and placing them into another empty container.
  Opening a loosely closed jar lid by gripping it with the help of the hand robot.
  Stacking checkers pieces on top of each other on an empty table. Picking up 5 cards from a table, flipping them over, and placing them back on the table.
  Grasping small weighted cubes from one table and transferring them to another table of a different height.
  These exercises were aimed at improving hand function and fine motor coordination.
  Interventions: Other: NDT+Hand Robot

INTERVENTIONS:
Other: NDT — The neurodevelopmental therapy program aimed to reduce muscle tone, improve hand functions, enhance fine motor skills, and support daily living activities such as eating and personal care.
  Specific exercises included:
  Finger and wrist flexion/extension, Shoulder and elbow stretching and mobilization, PNF exercises, Functional tasks like screw and nut manipulation, Velcro tasks, door handle turning, button pressing, zipper pulling, and laundry peg placement/removal.
  Arms: Neurodevelopmental Group
Other: NDT+Hand Robot — In this group, participants received 25 minutes of hand robot-assisted therapy following neurodevelopmental treatment. After the robot therapy, they performed fine motor skill exercises, including:
  Picking up buttons from one container and placing them in another, Opening a loosely closed jar lid using the robot, Stacking checkers pieces on a table, Flipping over and placing cards back on the table, Transferring weighted cubes from one table to another at a different height. These activities aimed to improve fine motor coordination and hand functionality.
  Arms: Hand Robot Group

SUMMARY:
This study aimed to evaluate the effectiveness of hand robot-assisted therapy on functionality, fine motor skills, and activities of daily living (ADLs) in acute stroke rehabilitation. A total of 30 participants aged 40-60 years with a diagnosis of stroke were randomly assigned to two groups: a neurodevelopmental treatment (NDT) group (n=15) and a hand robot-assisted therapy group (n=15). The NDT group received a standard rehabilitation program, including strengthening, stretching, and fine motor activities, three times per week for 8 weeks. The hand robot group received the same NDT program with the addition of hand robot therapy sessions three times per week for 8 weeks.

Outcome measures included the ABILHAND Stroke Questionnaire for hand function, the Barthel Index (BI) for ADLs, the Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire for functionality, the Nine-Hole Peg Test (NHPT) for fine motor skills, and the Modified Ashworth Scale (MAS) for spasticity. Both groups showed significant improvements in ADLs, fine motor skills, and ABILHAND scores after treatment (p<0.05). The hand robot group demonstrated superior improvements in BI and NHPT scores compared to the NDT group (p<0.05), while other parameters showed comparable results between groups.

Hand robot-assisted therapy may serve as a complementary approach to neurodevelopmental treatment in individuals with acute stroke.

DETAILED DESCRIPTION:
This study aimed to investigate the effectiveness of hand robot-assisted therapy on functionality, fine motor skills, and activities of daily living (ADLs) in individuals undergoing acute stroke rehabilitation. A total of 30 participants, aged 40-60 years and diagnosed with stroke, were randomly assigned into two groups: a neurodevelopmental treatment (NDT) group (n=15) and a hand robot-assisted therapy group (n=15).

The NDT group participated in a rehabilitation program consisting of strengthening, stretching, and fine motor activities, administered three times per week for 8 weeks. The hand robot-assisted therapy group received the same NDT program with the addition of hand robot therapy, performed three times per week for 8 weeks immediately after the NDT sessions.

Several assessment tools were used to evaluate outcomes: the ABILHAND Stroke Questionnaire for hand function, the Barthel Index (BI) for ADLs, the Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire for functionality, the Nine-Hole Peg Test (NHPT) for fine motor skills, and the Modified Ashworth Scale (MAS) for spasticity. Baseline characteristics, including age, sex, and stroke duration, were homogeneously distributed between groups.

Both groups exhibited significant improvements in ADLs, fine motor activities, ABILHAND scores, and NHPT results post-treatment compared to baseline (p<0.05). However, the hand robot-assisted therapy group demonstrated significantly greater improvements in BI and NHPT scores compared to the NDT group (p<0.05). For other parameters, both groups showed similar outcomes.

These findings suggest that hand robot-assisted therapy can be effectively utilized as a complementary approach to neurodevelopmental treatment in acute stroke rehabilitation, particularly in enhancing ADLs and fine motor skills.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 40-60 diagnosed with stroke
* Possession of adequate communication skills
* A score of at least 20 or higher on the Mini-Mental State Examination
* Full range of motion in the metacarpophalangeal (MCP), proximal interphalangeal (PIP), and distal interphalangeal (DIP) joints
* Spasticity score of 2 or below in the elbow, wrist, and finger flexor muscles according to the Modified Ashworth Scale
* Upper extremity muscle strength between 2+ and 4
* Stroke duration not exceeding 6 weeks

Exclusion Criteria:

* Inability to meet the study requirements due to insufficient verbal or written communication skills
* Presence of deformities that prevent participation in exercise
* Additional diagnoses of cardiovascular, rheumatologic, or orthopedic conditions
* Individuals who have undergone surgery within the past 6 months were excluded from the study

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-27 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-01-05 (Actual)

PRIMARY OUTCOMES:
Barthel Index | From enrollment to the end of treatment at 8 weeks
  The Barthel Index (BI) of Activities of Daily Living is used to assess participants' independence in performing daily activities without assistance. Scored between 0 and 100, the Barthel Index indicates total dependency in the range of 0-20 points, while a score of 100 represents complete independence.
ABILHAND | From enrollment to the end of treatment at 8 weeks
  In the study, the ABILHAND Stroke Hand Function Questionnaire, developed by Penta et al. was used to evaluate hand functions. The assessment examines the level of difficulty participants experience in performing daily tasks such as dressing, household chores, and eating. For the 56 tasks included in the questionnaire, participants are asked to rate their ability based on the past month using the following options: impossible (0 points), difficult (1 point), or easy (2 points) . A higher score indicates better hand function.
DASH | From enrollment to the end of treatment at 8 weeks
  The Disabilities of the Arm, Shoulder, and Hand (DASH) Questionnaire is used to assess physical limitations and function in upper extremity problems. The DASH questionnaire consists of three subparameters, with the first section comprising 30 questions. Of these, 21 questions evaluate the difficulties patients face in daily life functions, 5 questions assess symptoms, and the remaining 4 questions measure social function, work, sleep, and self-confidence levels.

SECONDARY OUTCOMES:
Nine Hole Peg Test | From enrollment to the end of treatment at 8 weeks
  The Nine-Hole Peg Test (NHPT), a timed test validated and reliable for stroke patients, was used to assess hand dexterity and fine motor skills. The test consists of a standard wooden block with 9 pegs (9 mm in diameter) and 9 holes (10 mm in diameter). Participants are instructed to pick up the pegs one by one and place them in the holes on the block as quickly as possible, then remove them individually. The time taken to insert and remove all pegs is recorded. The stopwatch starts when the participant first touches a peg and stops when the last peg is placed back on the table. Patients are allowed to stabilize the wooden block with their non-tested hand.
The Modified Ashworth Scale | From enrollment to the end of treatment at 8 weeks
  The Modified Ashworth Scale is the most commonly used method for assessing spasticity. The evaluation should be performed while the individual is lying supine in a relaxed position. The joint is moved passively, repeatedly, and rapidly, and the resistance felt during the movement is scored.

CONTACTS AND LOCATIONS:
Overall Officials: Burak Menek, Principal Investigator — Medipol University
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medipol University, Istanbul, Beykoz
  - NP Istanbul Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No